CLINICAL TRIAL: NCT03165188
Title: Long Term Follow-Up Study for Subjects Previously Treated With Algenpantucel-L (HyperAcute-Pancreas) Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: The IND was withdrawn
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Other Study IDs: NLG0705
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol (NLG0705) provides a mechanism for the 15-year follow-up period that the FDA requires for all participants in gene transfer protocols and assures that adequate follow-up can be maintained for subjects who have received at least one dose of algenpantucel-L.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of at least one dose of algenpantucel-L within the past 15 years
* Signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research subjects who have received at least one dose of algenpantucel-L immunotherapy in clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with adverse events. | Up to 15 years
Survival | Up to 15 years

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Cancer Center, Palo Alto, California
  - UF Health Cancer Center, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - University of Louisville, Louisville, Kentucky
  - Washington University, St Louis, Missouri
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Health Cancer Center, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided